CLINICAL TRIAL: NCT04697615
Title: Reliability of Algometry as a Clinical Value in Swimming Athletes
Brief Title: Reliability of Algometry in Swimming Athletes
Status: Completed | Type: Observational
Sponsor: São Paulo State University (Other)
Responsible Party: Sponsor
Other Study IDs: FIS190098
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Athletes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Algometry: In the test stage, pain threshold evaluations were started through the algometer in a randomized manner by two different examiners trained and experienced in the application of the test, following the same order of evaluation of the muscles (middle deltoid, upper trapezius, pectoralis major, biceps brachii , triceps, lumbar multifidus, rectus femoris, biceps femoris, tibialis anterior and soleus, bilaterally), with an interval between each assessment of five minutes in which the participants remained at rest. After the interval described, the retest stage was initiated, which had the same procedures as the test stage.
  Interventions: Device: Algometry

INTERVENTIONS:
Device: Algometry — The evaluation with the algometer was carried out in the same way by the two examiners, who held the instrument with the dominant hand, in order to adjust and coordinate the movements, while the non-dominant hand was used to stabilize the participant's skin, providing more security, avoiding thus small deviations. The pressure was applied at an angle of 90 ° (between the tool surface and the evaluated point), the rate of pressure increase was approximately 2 kg / cm² / s (kilogram per centimeter squared per second), up to the level that the participant reported a change in the sensation of pressure to a sensation of discomfort and immediately the examiner removed the device from the positioned location.

SUMMARY:
In the competitive swimming scenario, there is a significant incidence of pain, which can be justified by the high levels of training that exposes athletes to constant stress. In this way, the quantification of pain and its monitoring becomes extremely important for clinical practice. A commonly used tool with easy access and clinical applicability, capable of measuring the pain threshold (PT) in a standardized manner is the pressure algometer. However, there is a shortage in the literature of studies that evaluate the reliability of this instrument in healthy swimming athletes. Objectives: Evaluate the intra and inter-examiner reliability and to describe the profile of the PT measurements measured by the algometer in swimming athletes. Methods: It is a reliability study, and will be composed of fifty young athletes members of swimming teams, of both genders, aged between 12 and 20 years. The evaluation will be carried out on the same day and in 2 steps: (1) Test and (2) Retest. In the first step, through a third examiner, the participants will be subjected to marking of points in pre-determined muscles and in points of referred pain. Next, they will perform the PT assessment through the algometer by two other distinct and trained examiners. The interval between each examiner will be five minutes with the participant at rest. After five minutes the test was performed, the step retest will begin, which will have the same procedures as in the previous step. The statistical package SPSS Statistics 23.0 will be used to conduct the analyzes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy swimming athletes

Exclusion Criteria:

* Being an alcoholic and/or consuming drugs and/or smoking;
* Anti-inflammatory and / or analgesic drugs less than 24 hours before the test;
* Presenting anemia, inflammatory process, diabetes, cardiovascular disease;
* Episodes of muscle-tendon or osteoarticular injury in the lower, upper and / or lower limbs spine in the last three months;
* In addition to swimming for less than two years.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Young swimming athletes who regularly train and are members of the swimming teams of the 4th region of the state of São Paulo, of the São Paulo Aquatic Federation (FAP), of the cities of Presidente Prudente, Votuporanga and São José do Rio Preto.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Pain threshold | two hours
  Portable hand pressure algometer (FPX 50/220, Wagner Instruments, Greenwich, USA), measured in kg / cm² (kilogram per centimeter squared).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo State, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
Individual data will not be released, because participants are under eighteen.